CLINICAL TRIAL: NCT06010641
Title: Trendelenburg Position for Acute Anterior Circulation Ischemic Stroke With Large Artery Atherosclerosis Etiology (HOPES 3): a Prospective, Randomized, Open-label, Blinded-endpoint, Multi-center Trial
Brief Title: Trendelenburg Position for Acute Anterior Circulation Ischemic Stroke With Large Artery Atherosclerosis Etiology (HOPES 3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2023) 148
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head-down position (Experimental): head-down position as an adjunct to guideline-based treatment
  Interventions: Other: head-down position
- control (Other): guideline-based treatment
  Interventions: Other: head-down position

INTERVENTIONS:
Other: head-down position — -20° Trendelenburg as an adjunct to guideline-based treatment,

SUMMARY:
The effect of head position as a nonpharmacological therapy on acute ischemic stroke (AIS) remains inconclusive. Recent HOPES2 (Head dOwn-Position for acutE moderate ischemic Stroke with large artery atherosclerosis) suggest the safety, feasibility, and potential benefit of the head-down position (HDP) in acute ischemic stroke. The current study aims to investigate the efficacy and safety of HDP in acute moderate ischemic stroke patients with large artery atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Acute ischemic stroke confirmed by NCCT or MRI;
* Moderate neurologic deficit (6≤ NIHSS ≤ 16) within 24 hours of onset, or progressing from mild (NIHSS ≤ 5) to moderate neurologic deficit (6≤ NIHSS ≤ 16) within 24 hours, requiring ≥ 4 point increase in NIHSS score although the onset time is beyond 24 hours;
* Probable large artery atherosclerosis etiology based on the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria (responsible artery stenosis ≥ 50% or occlusion);
* Anterior circulation stroke (internal carotid artery, M1 or M2 of middle cerebral artery);
* First stroke onset or past stroke without obvious neurological deficit (mRS≤2);
* Signed informed consent.

Exclusion Criteria:

* Pre-stroke disability (mRS≥3);
* Patients with disturbance of consciousness;
* Patients who plan to undergo or have completed thrombolysis or mechanical thrombectomy;
* Hemorrhagic stroke or combined ischemic and hemorrhagic stroke;
* Serious comorbidity, such as liver or kidney insufficiency, malignant tumor, etc;
* Other stroke etiologies, such as cardiogenic embolism, arteritis, arterial dissection, moyamoya disease, etc;
* Previous history of intracerebral hemorrhage within 1 year;
* Any contraindication to head-down position (e.g. active vomiting, pneumonia, uncontrolled heart failure);
* Planned carotid or intracranial revascularization within 3 months;
* Severe uncontrolled hypertension (systolic blood pressure over 180mmHg or diastolic blood pressure over 100 mmHg);
* Cardiac insufficiency (NYHA Class ≥II);
* Pregnant or lactating women;
* Comorbidity with other serious diseases;
* Participating in other clinical trials within 3 months;
* Patients not suitable for the study considered by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
proportion of favorable functional outcome | 90±7 days
  favorable functional outcome defined as modified Rankin Score (mRS) 0-2. The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
proportion of excellent functional outcome | 90±7 days
  excellent functional outcome is defined as modified Rankin Score (mRS) 0-1. The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Score (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
early neurological deterioration (END) | 48±12 hours
  END is defined as more than 4-point increase in NIHSS within 48±12 hours, but was not a result of intracerebral hemorrhage
early neurological improvement (ENI) | 48±12 hours
  ENI is defined as more than 4-point decrease in NIHSS within 48±12 hours
Changes in National Institute of Health stroke scale (NIHSS) | 48±12 hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
Changes in National Institute of Health stroke scale (NIHSS) | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
changes in infarct volume | 48±12 hours
new stroke or other vascular event(s) | 90±7 days
all-cause mortality | 90±7 days

OTHER OUTCOMES:
changes in cortical oxygen saturation determined by near infrared spectroscopy | 24±8 hours
changes in cortical oxygen saturation determined by near infrared spectroscopy | 48±12 hours
changes in serum biomarkers | 48±12 hours
changes in serum biomarkers | 10±2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li X, Guo Z, Wang L, Wang Y, Nguyen T, Yang Y, Chen HS. Trendelenburg position for acute anterior circulation ischaemic stroke with large artery atherosclerosis aetiology (HOPES 3): rationale and design. Stroke Vasc Neurol. 2024 Nov 5;9(5):574-579. doi: 10.1136/svn-2023-002868. PMID 38296589